CLINICAL TRIAL: NCT01607827
Title: Colorectal Polypectomy Upon Insertion And Withdrawal Or Upon Withdrawal Only?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Stephan Wildi, Stephan M. Wildi, Principle Investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EK-1066
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Polyps
Keywords: polypectomy; colonoscopy; polyp miss rate; surveillance; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyp removal upon insertion and withdrawal (Active Comparator)
  Interventions: Procedure: Polyp removal upon insertion and withdrawal
- Polyp removal upon withdrawal only (No Intervention)
  Interventions: Procedure: Polyp removal upon withdrawal only

INTERVENTIONS:
Procedure: Polyp removal upon insertion and withdrawal — Endoscopic procedures:
  All polypectomies in the study groups were performed using the same techniques as in the standard care of non-study patients, using snare loops, hot biopsy forceps, with and without submucosal injection of saline/epinephrine. Polyps larger than 3 mm were removed by snare, polyps smaller than 4 mm were removed by cold biopsy. There were no differences upon insertion or withdrawal.
  The endoscopist removed all visible polyps instantly regardless whether advancing the instrument to the cecum or pulling back.
  Arms: Polyp removal upon insertion and withdrawal
Procedure: Polyp removal upon withdrawal only — Endoscopic procedures:
  All polypectomies in the study groups were performed using the same techniques as in the standard care of non-study patients, using snare loops, hot biopsy forceps, with and without submucosal injection of saline/epinephrine. Polyps larger than 3 mm were removed by snare, polyps smaller than 4 mm were removed by cold biopsy. There were no differences upon insertion or withdrawal.
  The endoscopist advanced the endoscope to the cecum without removing polyps. Upon withdrawal, all visible polyps were removed successively by standard techniques.
  Arms: Polyp removal upon withdrawal only

SUMMARY:
The investigators aim to assess the procedure time and miss rate of polyps when performing polypectomy in the colon on the way up* and down** or only on the way down**.

(* advancing the scope to the cecum, ** pulling back the scope after intubation of the cecum). Our hypothesis is that using the strategy to remove all visible polyps firstly on the way up and secondly on the way down is less time consuming and misses less polyps as with the strategy to remove polyps only on the way down.

DETAILED DESCRIPTION:
Patients with a referral for a complete colonoscopy were included in the study. Polyps were removed upon insertion and withdrawal of the colonoscope in Group A or only upon withdrawal of the instrument in Group B according to a computer-generated randomization list.

The following inclusion criteria were used: referral for a complete colonoscopy and age of 18 years and older. All patients with polyps detected during colonoscopy were included. In order to compare the time required for the entire endoscopy between the two treatment groups, we only included patients with polyps of up to 10 mm in diameter.

The following exclusion criteria were applied: colonoscopy due to bleeding, high likelihood of colonic stenosis or severe inflammation, inflammatory bowel disease (IBD), hereditary colonic polyp disease (FAP or HNPCC), contraindications for polypectomy, such as coagulopathy, use of anti-clotting medication (anticoagulation, high-dose heparin aspirin, NSAIDs), polyps >10 mm in diameter (that cannot be removed through the biopsy channel and have to be removed by basket or polyp grasper; the use of these devices necessitates removal and consecutive re-insertion of the endoscope, making a comparison of the time intervals between the two groups impossible), suboptimal bowel preparation (presence of significant amounts of fecal remnants that could not be removed by flushing of the colon over the colonoscope and that did not allow clear visualization of the mucosa), and missing signed informed consent form.

The randomization was done as soon as the first polyp was detected. When no polyps were detected, the case was regarded as screening failure and excluded from the study.

Randomization was performed into the following two groups:

Group A: Removal of all visible polyps upon insertion and withdrawal of the instrument Group B: Removal of all visible polyps upon withdrawal of the colonoscope only One day after colonoscopy, patients were asked to complete a questionnaire evaluating the tolerance of the ileo-colonoscopy (on a visual scale from 1 to 4 where 1 stands for no discomfort, 2 for minor discomfort, 3 for moderate discomfort, and 4 for severe discomfort associated with the endoscopy).

Endoscopic procedures:

Colon preparation was performed using 3 liters of PEG-based standard lavage fluids (Fordtran Streuli ®, Streuli Pharma, Switzerland).

The procedures were performed by senior endoscopists (SW, SRV, HF, NW, PB) with at least 5 years of experience in colonoscopy and performing at least 200 colonoscopies per year. All endoscopists participating in this trial underwent a specific study training headed by SW. Polyp size was measured using an opened biopsy forceps (Boston Scientific Radial JawTM 4, Reference No 1332, diameter of opened jaws 9mm). All endoscopists had comparable numbers of procedures in both approaches to polypectomy.

Premedication consisted mostly of propofol (60-400 mg) or a combination of midazolam (2.5-5 mg) and/or meperidine (25-50 mg) intravenously. Examinations were performed in left lateral decubitus or supine position. Colonic insufflation was performed with room air. All polypectomies in the study groups were performed using the same techniques as in the standard care of non-study patients, using snare loops, hot biopsy forceps, with and without submucosal injection of saline/epinephrine. Polyps larger than 3 mm were removed by snare, polyps smaller than 4 mm were removed by cold biopsy. There were no differences upon insertion or withdrawal.

In Group A, the endoscopist removed all visible polyps instantly regardless whether advancing the instrument to the cecum or pulling back. In Group B, the endoscopist advanced the endoscope to the cecum without removing polyps. Upon withdrawal, all visible polyps were removed successively by standard techniques. In both groups, the endoscopists were instructed to focus on rapid introduction.

Assessments After the endoscopy, the physician completed the data capture sheet evaluating the following criteria: patient demographics, patient history, time intervals required for the procedure, number of polyps detected upon insertion, number of polyps removed upon insertion, number of polyps removed upon withdrawal, overall technical ease (score from 1 to 4 where 1 stands for no technical problems, 2 for minor, 3 for moderate, and 4 for major technical difficulties), presence of technical problems (difficult visualization of the polyps, difficult removal of polyps, and difficult retrieval of polyps, all answered categorically with "Yes" or "No"), patient tolerance (completed by patients), and characterization of every polyp (location, size, time of removal and additional comments).

ELIGIBILITY:
Inclusion Criteria:

* Need for a complete colonoscopy
* 18 years of age and older

Exclusion Criteria:

* Need for urgent colonoscopy due to bleeding
* High likelihood of colonic stenosis or severe inflammation
* Known inflammatory bowel disease (IBD)
* Known familiarity adenomatous polyposis (FAP)
* Contraindications for polypectomy such as coagulopathy, use of anti-clotting medication (anticoagulation, aspirin, NSAIDs)
* Missing signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-04; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Polyp detection | 2004 - 2007

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M. Wildi, MD, Principal Investigator — University of Zurich
Locations (1):
- University of Zürich, Zurich, Canton of Zurich, Switzerland